CLINICAL TRIAL: NCT02574611
Title: Safety and Efficacy of High Resolution Manometry in Studying Colonic Motility and Iontophoretic Administration of Prokinetic Agents
Brief Title: Use of High Resolution Colonic Manometry in Studying Motility
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No reportable findings are possible. The PI/Co-PI were unable to recruit participants for this study. One participant was consented but did not undergo any study procedure.
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Mark Korsten, Chief Gastroenterologist, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: KOR-15-026
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Dysfunction
MeSH Terms: interventions — Neostigmine; Glycopyrrolate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- SCI observational (Experimental): Individuals with SCI will undergo a one day observation following elective colonoscopy and placement of the colonic catheter. Investigators will be monitoring colonic motility during a "typical" day (eating, sleeping, mobility, etc.).
  Interventions: Device: High Resolution Colonic Manometry
- Able-bodied observational (Experimental): Able-bodied individuals (non SCI) will undergo a one day observation following elective colonoscopy and placement of the colonic catheter. Investigators will be monitoring colonic motility during a "typical" day (eating, sleeping, mobility, etc.).
  Interventions: Device: High Resolution Colonic Manometry
- SCI drug group (Active Comparator): Individuals with SCI will undergo a second day observation following elective colonoscopy and placement of the colonic catheter. Investigators will be monitoring colonic motility during the transdermal administration of neostigmine and glycopyrrolate.
  Interventions: Drug: Neostigmine; Drug: Glycopyrrolate; Device: High Resolution Colonic Manometry
- SCI placebo group (Placebo Comparator): Individuals with SCI will undergo a second day of observation following elective colonoscopy and placement of the colonic catheter. Investigators will be monitoring colonic motility during the transdermal administration of normal saline solution (placebo).
  Interventions: Other: Saline (Placebo); Device: High Resolution Colonic Manometry

INTERVENTIONS:
Drug: Neostigmine
  Arms: SCI drug group
Drug: Glycopyrrolate
  Arms: SCI drug group
Other: Saline (Placebo)
  Arms: SCI placebo group
Device: High Resolution Colonic Manometry

SUMMARY:
An injury to the spinal cord (SCI) results in numerous medical complications, including gastrointestinal (GI) function. Individuals with SCI may experience severe constipation (prolonged stool retention), incontinence (accidents), and overall difficulty in bowel evacuation. While various treatments and medications have been established to address this complication, there is little knowledge relating to the overall colonic motility. However, new technology such as High Resolution Colonic Manometry allows physicians to visualize high pressure contractions inside the colon, leading to a greater understanding of typical motility, a more accurate diagnosis, and an effective treatment. In this study, the investigators propose to use this technology to understand the effects of SCI on colonic motility by comparing to normal colonic function observed in able-bodied (AB) individuals. In addition, the investigators plan to study the effects of pharmacological treatments, such as neostigmine, on promoting peristaltic contractions in the colon as it is delivered across the skin.

DETAILED DESCRIPTION:
The investigators data suggests that the fundamental consequence of SCI is a slowing of intestinal peristaltic activity, most likely as a result of down regulation of parasympathetic neural pathways. Furthermore, the investigators have effectively shown that measures involved in increase parasympathetic stimulation results in efficient bowel evacuation and improved bowel care. Such measures include the administration of neostigmine (NEO), which increases peristaltic contractions in the colon, resulting in predictable bowel evacuations. Given the cardiopulmonary side-effects of NEO, an ant-cholinergic known as Glycopyrrolate (GLY) is usually co-administered with NEO to reverse these side effects. However, the investigators knowledge regarding the effects of SCI on colonic motility is still primitive, mainly due to pervious technological disadvantages. New High Resolution Colonic Manometry systems (Medical Measurement Systems Dover, NH) simultaneously capture high amplitude pressure contractions (HAPCs) across the ascending, transverse, descending, and recto-sigmoid colon. Such capabilities allow for a much clearer display of pressure events compared to previous line tracing manometric systems and the direction of contractions are much easier to discern as well. To date, this technology has been an effective tool in diagnosing bowel disorders and complications, such as constipation in able-bodied individuals (AB). However, such studies have not been conducted in a SCI population. This technology also has the potential to capture the effects of NEO+GLY on improving colonic function.

ELIGIBILITY:
Inclusion Criteria:

* Chronic SCI >1year
* Able-Bodied (non SCI)
* Undergoing Elective Colonoscopy
* Age 18-75 years.

Exclusion Criteria:

* Previous adverse reaction or hypersensitivity to electrical stimulation
* Known sensitivity to neostigmine or glycopyrrolate
* Persons with SCI who do not require additional bowel care or have "normal bowel function"
* Known hypersensitivity to neostigmine or glycopyrrolate
* History of mechanical obstruction of the intestine or urinary tract
* History of Myocardial infarction
* Uncontrollable Hypertension Defined by a blood pressure reading of 160/100 mmHg or higher
* Organ damage (heart & kidney) and/or transient ischemic attack-cerebral vascular accident as a result of hypertension
* Known past history of coronary artery disease or bradyarrythmia
* Active respiratory disease
* Known history of asthma during lifetime or recent (within 3 months) respiratory infections
* Adrenal insufficiency
* Diagnosed coagulopathy
* Any renal disease or dysfunction
* Potential for pregnancy
* Lactating/nursing females
* Slow-heart beat (HR<45 bpm)
* Lack of mental capacity to give consent
* Use of any antibiotic in the past 7 days
* Use of medications known to affect the respiratory system
* Use of medications known to alter airway caliber
* Concurrent participation in other clinical trials (within 30 days)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
High Amplitude Contractions | 1-2days
  Monitor changes in High Amplitude Contractions inside the colon during a typical day for SCI and AB patients. The manometry system will record these changes and allow the investigators to visualize changes during various activities (eating, resting, supine, seated, walking, etc.) The investigators will also measure changes in contractions during administration of prokinetic agents to promote bowel evacuations

CONTACTS AND LOCATIONS:
Overall Officials: Mark Korsten, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No